CLINICAL TRIAL: NCT01623414
Title: Sunlight Exposure and Vitamin D Status of Children of South Asian Ethnicity Living in the UK
Status: Completed | Type: Observational
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Lesley Rhodes, Professor of Experimental Dermatology, University of Manchester
Other Study IDs: AMR-1950
Record Dates: First submitted 2012-06-13; First posted 2012-06-20 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy schoolchildren

SUMMARY:
The purpose of this study is to examine the amount of sunlight exposure and vitamin D status of adolescent schoolchildren of South Asian ethnicity in each season throughout the year.

ELIGIBILITY:
Inclusion Criteria:

* Healthy schoolchildren aged 12-15 years
* Sun-reactive skin type V (naturally brown skin)
* South Asian ethnicity
* Male or female

Exclusion Criteria:

* History of photosensitivity disorder
* Non-ambulant

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Schoolchildren of South Asian ethnicity in Greater Manchester
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2012-09; Primary Completion 2013-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change in serum concentration of 25-hydroxyvitamin D | 1 year
  Serum vitamin D will be assessed every 3 months over a period of 1 year

SECONDARY OUTCOMES:
Change in sunlight exposure received | 1 year
  Exposure to sunlight over 7 consecutive days is measured using polysulphone badges with one badge for weekdays and a second badge for the weekend. Exposure is assessed every 3 months for 1 year.
Change in dietary intake of vitamin D | 1 year
  Intake of foods containing vitamin D is recorded for a one week period once every 3 months over a period of 1 year and the average daily intake determined.

CONTACTS AND LOCATIONS:
Overall Officials: Lesley Rhodes, MD FRCP(UK), Principal Investigator — University of Manchester
Locations (1):
- Salford Royal NHS Foundation Trust, Manchester, United Kingdom